CLINICAL TRIAL: NCT02978248
Title: Af Register RhEin NeckAr - Projekt Vorhofflimmern Rhein Neckar
Brief Title: ARENA - Project Atrial Fibrilation Rhine-Neckar Region
Acronym: ARENA
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: ARENA
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
ARENA aims to inform patients about the symptoms and the risks of atrial fibrilation.

The study design includes three study arms:

1. ARENA Intervention: This project will examine the effectiveness of population education.
2. ARENA Medication: The aim is to examine the patient's adherence and to analyze whether there are any complications.
3. ARENA Migration: ARENA migration aims to examine whether a targeted population education can improve the care of people with a Turkish migration background.

DETAILED DESCRIPTION:
ARENA aims to inform patients about the symptoms and the risks of atrial fibrilation.

The study design includes three study arms:

1. ARENA Intervention:

   This project will examine the effectiveness of population education and other measures to provide care for patients with atrial fibrillation.

   In the end of the control phase (1 year recruitment of approximately 10,000 patients), there will be a wide publicity, informing about the disease.
2. ARENA Medication:

   ARENA records the patient's complete medication at all survey times (up to two weeks after recruitment and follow up). This allows an accurate assessment of interactions between individual substances.

   In addition, attempts are being made to determine drug concentrations of anticoagulants directly by the blood of the patient. Therefore, patients are provided with kits, which they can use to apply a drop of blood from your fingertip to a filter paper. The aim is to examine the patient's adherence and to analyze whether there are any complications.
3. ARENA Migration:

The Metropolregion Rhein-Neckar is characterized by a high proportion of people with a Turkish migration background. ARENA migration aims to examine whether a targeted population education can improve the care of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Atiral fibrilation
* 18 years or older

Exclusion Criteria:

* Not willing to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrilation in the Rhein-Neckar Region in Germany, recruted by their general practitioner or during a hospital stay.
Sampling Method: Probability Sample
Enrollment: 2777 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Number of Prevented strokes in participants | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Borggrefe, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim; Walter E. Haefeli, Prof. Dr., Study Chair — University Hospital Heidelberg; Ömer Sanatci, Dr. med., Study Chair — Praxis Merz Sanatci
Locations (1):
- Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brockmuller C, Meid AD, Senges J, Hochadel M, Haefeli WE, Stoll F. Phenotypes of Patients with Direct Oral Anticoagulant (DOAC) Underdosing in Atrial Fibrillation: Results from the ARENA Registry. Clin Drug Investig. 2025 Jan;45(1):29-43. doi: 10.1007/s40261-024-01411-w. Epub 2024 Dec 12. PMID 39666256
- [Derived] Zylla MM, Ozdemir B, Hochadel M, Zeymer U, Akin I, Grau A, Schneider S, Alonso A, Waldecker B, Suselbeck T, Schwacke H, Haass M, Zahn R, Borggrefe M, Senges J, Frey N, Thomas D. Community-based analysis of stroke prevention and effect of public interventions in atrial fibrillation: results from the ARENA project. Clin Res Cardiol. 2025 Jan;114(1):138-149. doi: 10.1007/s00392-024-02510-6. Epub 2024 Aug 8. PMID 39115608
- [Derived] Sadlonova M, Salzmann S, Senges J, Celano CM, Huffman JC, Borggrefe M, Akin I, Thomas D, Schwarzbach CJ, Kleemann T, Schneider S, Hochadel M, Suselbeck T, Schwacke H, Alonso A, Haass M, Ladwig KH, Herrmann-Lingen C. Generalized anxiety is a predictor of impaired quality of life in patients with atrial fibrillation: Findings from the prospective observational ARENA study. J Psychosom Res. 2024 Jan;176:111542. doi: 10.1016/j.jpsychores.2023.111542. Epub 2023 Nov 8. PMID 37977094